CLINICAL TRIAL: NCT00695201
Title: A Phase I Study of Hepatic Arterial Infusion With Floxuridine and Dexamethasone in Combination With Intravenous Oxaliplatin Plus Irinotecan in Patients With Unresectable Hepatic Metastases From Colorectal Cancer.
Brief Title: Hepatic Arterial Infusion With Floxuridine and Dexamethasone in Combination With Intravenous Oxaliplatin Plus Irinotecan in Patients With Unresectable Hepatic Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Medicine and Dentistry of New Jersey (Other); Rutgers, The State University of New Jersey (Other); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-011
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: DEXAMETHASONE; FLOXURIDINE; IRINOTECAN (CPT-11) CAMPTOSAR; OXALIPLATIN
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Floxuridine; Oxaliplatin; Irinotecan

ARMS (2):
- 1 (Experimental): Patients will undergo pump placement and biopsy of diseased liver tissue. Chemotherapy will be initiated as soon as possible following verification of adequate pump placement and perfusion by radiographic pump study. Treatment will continue indefinitely unless a patient experiences a treatment endpoint.
  Interventions: Drug: Floxuridine, Oxaliplatin, CPT-11
- 2 (Experimental): Patients will undergo pump placement and biopsy of diseased liver tissue. Chemotherapy will be initiated as soon as possible following verification of adequate pump placement and perfusion by radiographic pump study. Treatment will continue indefinitely unless a patient experiences a treatment endpoint.
  Interventions: Drug: Floxuridine, Oxaliplatin, CPT-11

INTERVENTIONS:
Drug: Floxuridine, Oxaliplatin, CPT-11 — For patients on the 4-week cycle: On the first day of each cycle, the pump will be filled with FUDR and dexamethasone. The pump will be emptied of drugs after 2 weeks (on day 15 of each cycle) and filled with heparin (which is used to prevent blood from clotting) and saline. Whether the pump contains drug or heparin and saline, it will need to be emptied and refilled about every two weeks. We will inject either the drugs or the saline and heparin into the pump through the skin using a needle and syringe. In summary, 2 weeks of drug in the pump is followed by 2 weeks without drug in the pump. The systemic chemotherapy (Oxaliplatin/CPT-11) will be administered on the same day as the pump is filled and emptied, ie. Day 1 and Day 15 of each cycle.
  Arms: 1
Drug: Floxuridine, Oxaliplatin, CPT-11 — For patients on the 5-week cycle: On the first day of each cycle, the pump will be filled with FUDR and dexamethasone. The pump will be emptied of drugs after 2 weeks (on day 15 of each cycle) and filled with heparin and saline. This is repeated on day 29 of each cycle). In summary, 2 weeks of drug in the pump are followed by 3 weeks without drug in the pump. The systemic chemotherapy (Oxaliplatin/CPT-11) will be administered on the same day that the pump is emptied and filled with heparin and saline, i.e. Day 15 and Day 29 of each cycle.
  Arms: 2

SUMMARY:
The purpose of this study is to see how well patients tolerate the side effects of treatment with Floxuridine, Oxaliplatin and Irinotecan. We also want to know if these methods used together are a useful way of treating cancer. We have studied these drugs and know the best doses of each when they are used alone. We do not yet know how well the drugs work with each other. This study will tell us the best doses of each drug when they are given over the same period of time.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed colorectal adenocarcinoma metastatic to the liver with no clinical or radiographic evidence of extrahepatic disease.

Confirmation of diagnosis must be performed at MSKCC.

* Patient's liver metastases must be deemed unresectable and comprise <70% of the liver parenchyma.
* A patient may have had prior chemotherapy or be previously untreated.
* Patient may not have received prior treatment with FUDR or >2 doses of Oxaliplatin.
* KPS > or = to 60%.
* WBC > or = to 3,000 cells/mm3 and platelet count > or = to 100,000 cells/mm3 within 14 days of registration.
* Creatinine < or = to 1.5 mg/dl within 14 days of registration.
* Total serum bilirubin < or = 2.0 mg/dl within 14 days of registration.

Exclusion Criteria:

* No active concurrent malignancies: except a patient's potentially resectable colorectal primary.
* Patient must not have obstruction of GI or GU tract.
* Patient must not have current, symptomatic peripheral sensory neuropathy.
* No prior radiation to liver.
* No active infection, ascites, or hepatic encephalopathy.
* Age ≥ 18 years.
* Female patients cannot be pregnant or lactating.
* Signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2000-08; Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Determine the MTD of hepatic arterial floxuridine (FUDR) & dexamethasone (Dex) given via implanted pump in combination w biweekly intravenous Oxaliplatin + systemic irinotecan (CPT-11) in patients w unresectable hepatic metastases from colorectal cancer. | conclusion of the study

SECONDARY OUTCOMES:
To determine the preliminary anti-tumor activity of the aforementioned combination chemotherapy. | conclusion of the study
To procure normal and disease liver tissue for evaluation of TS, p53, p21, TOPO 1, DPD, and ERCC levels. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kemeny, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org